CLINICAL TRIAL: NCT00168129
Title: Helical Tomotherapy as a Radiotherapy Technique for Treating Bone Metastases
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alberta Health services (Other)
Organization: AHS Cancer Control Alberta (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA-15-0007
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2011-12-09 (Estimated); Status verified 2011-12

CONDITIONS: Bone Neoplasms
Keywords: tomotherapy; bone metastases; radiotherapy; intensity modulated
MeSH Terms: conditions — Bone Neoplasms | interventions — Radiotherapy, Intensity-Modulated

INTERVENTIONS:
Procedure: Helical tomotherapy

SUMMARY:
To assess the safety and efficacy of a single fraction of radiotherapy using helical tomotherapy to treat bone metastases.

ELIGIBILITY:
Inclusion Criteria:

* painful metastatic bone disease from any malignancy

Exclusion Criteria:

* previous RT to same area
* contraindications to RT

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10
Dates: Start 2001-06; Study Completion 2005-07

PRIMARY OUTCOMES:
To deliver a single fraction of radiotherapy safely to patients with bone metastases using helical tomotherapy

SECONDARY OUTCOMES:
To assess and quantify the acute toxicity of patients with bone metastases treated with helical tomotherapy.
To measure invivo dosimetry and compare delivered doses to computer-reconstructed dose distribution.
To determine the maximum tolerated does of palliative radiation give with helical tomotherapy in a single fraction.
To assess the efficacy (pain control) of radiotherapy given with helical tomotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Rufus Scrimger, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada